CLINICAL TRIAL: NCT01069185
Title: Differences in Morbidity Frequency Between a Necessity Endotracheal Suctioning Protocol Versus a Routine Endotracheal Suctioning Protocol in Hospital Pablo Tobon Uribe´s Pediatric Intensive Care Unit (PICU). A Randomized Controlled Trial
Brief Title: Differences in Morbidity Between a Necessity Endotracheal Suctioning Protocol Versus a Routine Endotracheal Suctioning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Pablo Tobón Uribe (Other)
Responsible Party: Principal Investigator, Gloria Lema, MD, Hospital Pablo Tobón Uribe
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5100-66779
Record Dates: First submitted 2010-02-10; First posted 2010-02-17 (Estimated); Results first posted 2017-09-11 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Hypoxemia; Arrhythmias; Cardiac Arrest; Ventilator Associated Pneumonia
Keywords: Unplanned extubation; Length of stay in PICU; Length of mechanical ventilation
MeSH Terms: conditions — Hypoxia; Arrhythmias, Cardiac; Heart Arrest; Pneumonia, Ventilator-Associated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Necessity endotracheal suctioning (Experimental): Endotracheal suctioning depends on clinical manifestations
  Interventions: Procedure: Necessity endotracheal suctioning
- Routine endotracheal suctioning (Other): Endotracheal suctioning every two hours
  Interventions: Procedure: Routine endotracheal suctioning

INTERVENTIONS:
Procedure: Necessity endotracheal suctioning — Endotracheal suctioning depends on clinical manifestations
  Arms: Necessity endotracheal suctioning
Procedure: Routine endotracheal suctioning — Endotracheal suctioning every two hours
  Arms: Routine endotracheal suctioning

SUMMARY:
Morbidity frequency associated to a endotracheal suctioning is different between a necessity endotracheal suctioning protocol versus a routine endotracheal protocol.

DETAILED DESCRIPTION:
Endotracheal aspiration is a very useful procedure. It has several adverse events every time that aspiration is practiced. This trials wants to identify which protocol (necessity versus routine) could be better to practice in pediatrics intensive care unit with less risk.

ELIGIBILITY:
Inclusion Criteria:

* Children older than 1 month until 14 years old requiring orotracheal intubation

Exclusion Criteria:

* High frequency ventilation mode

Ages: 1 Month to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2010-02; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gloria L Lema, MD, Principal Investigator — Hospital Pablo Tobon Uribe
Locations (1):
- Hospital Pablo Tobon Uribe, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lema-Zuluaga GL, Fernandez-Laverde M, Correa-Varela AM, Zuleta-Tobon JJ. As-needed endotracheal suctioning protocol vs a routine endotracheal suctioning in Pediatric Intensive Care Unit: A randomized controlled trial. Colomb Med (Cali). 2018 Jun 30;49(2):148-153. doi: 10.25100/cm.v49i2.2273. PMID 30104806

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Necessity Endotracheal Suctioning | Routine Endotracheal Suctioning
Started | 47 | 45
Completed | 47 | 45
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Units Other Than Participants: suctioning number
Groups:
- Total: Total of all reporting groups
Arm/Group | Necessity Endotracheal Suctioning | Routine Endotracheal Suctioning | Total
Number analyzed (Participants) | 47 | 45 | 92
Number analyzed (suctioning number) | 606 | 649 | 1255
Age, Continuous [Median (Inter-Quartile Range); unit: months] | 34 [7 to 104] | 56 [14 to 108] | 40.5 [8.3 to 107.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 23 | 44
  Male | 26 | 22 | 48
Weight [Median (Inter-Quartile Range); unit: Kgs] | 15 [7 to 31] | 15 [10 to 30] | 15 [7.6 to 30]
PRISM [Median (Inter-Quartile Range); unit: units on a scale] — The PRISM score predicts the risk of mortality in critical children. It evaluates the degree of severity of the illness. Ranges are established between 0-100. As highest the number as highest the probability of dead.
  units on a scale | 23 [14 to 28] | 23 [17 to 27] | 23 [15 to 26.5]

OUTCOME MEASURES:

1. Primary Outcome: Primary Composite End Point
Description: All causes of morbidity. Clinically identified as hypoxaemia, unplanned extubation, cardiac arrythmias, cardiac arrest. Measured as any change in patient´s monitor identified for ancillary nurse and/or confirmed directly by pediatrician.
Time Frame: Every component for primary outcome can be assessed during or after suctioning is applied.For routine protocol, every 2 hours for necessity protocol will depend on patient´s necessity. The assessment was done in each patient during intubation period .
Measure: Number; unit: event
Units Other Than Participants: suctioning
Arm/Group | Necessity Endotracheal Suctioning | Routine Endotracheal Suctioning
Number analyzed (Participants) | 47 | 45
Number analyzed (suctioning) | 606 | 649
event | 35 | 48

2. Secondary Outcome: Mechanical Ventilation Length as Days.
Description: Number of days under mechanical ventilation during ICU hospitalization length
Time Frame: Every day while patient really is intubated.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Necessity Endotracheal Suctioning | Routine Endotracheal Suctioning
Number analyzed (Participants) | 47 | 45
Days | 2.5 [1 to 5] | 2.4 [0.8 to 6.4]

ADVERSE EVENTS:
Arm/Group | Necessity Endotracheal Suctioning | Routine Endotracheal Suctioning
All-Cause Mortality (participants affected / at risk) | 9/47 | 12/45
Serious Adverse Events (participants affected / at risk) | 0/47 | 1/45
Other Adverse Events (participants affected / at risk) | 0/45 | 0/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Necessity Endotracheal Suctioning (N=47) | Routine Endotracheal Suctioning (N=45)
VAP (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Ventilator Associated Pneumonia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes